CLINICAL TRIAL: NCT06349785
Title: Effect of Combined Manual Hyperinflation and Standard Physical Therapy Program on Lung Recruitment in Mechanically Ventilated Pediatric Patients: A Randomized Clinical Trial
Brief Title: Manual Hyperinflation and Physical Therapy Program on Lung Recruitment Mechanically Ventilated Pediatric Patients
Acronym: MHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Lecturer of Physical Therapy for Pediatrics and its Surgeries, New Ismailia National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/003858
Record Dates: First submitted 2024-03-23; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation Complication; Physical Disability
Keywords: MHI, Physical Therapy, Mechanically ventilated patients
MeSH Terms: interventions — Palliative Care; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: using sealed envelopes,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group A (Experimental): Assigned Children in the study will receive manual hyperinflation and standard physical therapy program. Manual hyperinflation (MHI): Manual hyperinflation will be performed by single physical therapist using a silicone resuscitator bag . The resuscitator bag (maximum volume of 500 mL) was connected to a pressure manometer with an oxygen flow of 10 L. min-1 with the total duration of session in group A will be 15 minutes, daily for 2 weeks
  Interventions: Device: rehabilitation of mechanically ventilated patients; Procedure: supportive care
- study group B (Active Comparator): - Children in study group B will receive standard Physical therapy program including suction, percussion and vibration with total duration of session in group a will be 15 minutes, daily for 2 weeks
  Interventions: Procedure: supportive care

INTERVENTIONS:
Device: rehabilitation of mechanically ventilated patients — 1. mechanical ventilation
  2. silicon resuscitation bag (500ml) connected to pressure manometer with an oxygen flow of 10 l.min-1
  3. Endotracheal closed suction with pressure control ventilation (PCV)
  Other Names: rehabilitation by using combined physical therapy and manual hyperinflation
  Arms: study group A
Procedure: supportive care — - Children in study group B will receive standard Physical therapy program including suction, percussion and vibration with total duration of session in group a will be 15 minutes, daily for successive two weeks
  Other Names: physical therapy for pediatric respiratory disorders

SUMMARY:
The purpose of this study is to investigate the immediate combined effects of Manual Hyperinflation and standard Physical therapy program on lung recruitment and secretion mass in mechanically ventilated pediatric patients aged between 10-15 years 'old

DETAILED DESCRIPTION:
In developing countries, lower respiratory tract infection is a major cause of death in children, with severely ill patients being admitted to the critical-care unit. While physical therapists commonly use the manual hyperinflation (MHI) technique for secretion mass clearance in critical-care patients, its efficacy has not been determined in pediatric patients.

Manual hyperinflation is a frequently maneuver used in critically ill intubated and mechanically ventilated patients. With MHI, patients are disconnected from the mechanical ventilator after which their lungs are temporarily ventilated with a manual ventilation bag. so, by applying a larger than normal volume at a low inspiratory pause and expiration with a high expiratory flow, MHI is suggested to mimic a normal cough.

Propagation of airway secretions from the smaller toward the larger airways, then allows for easy removed of airway secretions with the airway suction. finally, MHI could prevent airway plugging and even promote alveolar recruitment. so the aim of the study is to enhance lung recruitment using MHI combined with standard Physical therapy program

ELIGIBILITY:
Inclusion Criteria:

* The patients will be aged 10-15 years,
* receiving mechanical ventilation via an endotracheal tube for at least 24 h
* presenting with vital signs in the normal range.
* All patients are suffering from lower respiratory tract infection like pneumonia, bronchitis and acute exacerbation of bronchiectasis

Exclusion Criteria:

* Patients with history of thoracic surgery
* Patients with pneumothorax or acute respiratory distress syndrome
* Patients with severe acute head injury
* Patients use inotropes and vasopressors drugs
* Patients with severe Broncho pleural fistula, rib fracture, emphysema bullae, lung abscess, patients with history of preterm birth or heart disease.
* Patients who requiring mechanical ventilation with a peak inspiratory pressure (PIP)

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
change the respiratory functions | 2 weeks
  By increasing tidal volume
change the respiratory mechanics | 2 weeks
  increasing inspiratory capacity
change the bronchospasm | 2 weeks
  modifying mean airway pressure
change the amount of ventilation | 2 weeks
  increasing the oxygen saturation

SECONDARY OUTCOMES:
decreasing the amount of secretions | 2 weeks
  by monitoring the change of amount of secretions collection calibrated tube attached to a closed suction system to calculate the secretion mass before and after treatment using: Suction by Endotracheal closed suction with pressure control ventilation (PCV) will be performed. The duration of suction was 10 s with 5-s rest for each set. Three sets of suction with a closed suction system will be used for both groups of patients.
weaning from mechanical ventilator | from 2 to 4 weeks
  by improving previously mentioned respiratory function

CONTACTS AND LOCATIONS:
Overall Officials: Amr K Abo Takia, MD, Study Director — college of medicine Suez Canal University
Locations (1):
- College of Medicine, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
data will not be available to other researchers

REFERENCES:
- [Background] Ubeda Tikkanen A, Nathan M, Sleeper LA, Flavin M, Lewis A, Nimec D, Mayer JE, Del Nido P. Predictors of Postoperative Rehabilitation Therapy Following Congenital Heart Surgery. J Am Heart Assoc. 2018 May 12;7(10):e008094. doi: 10.1161/JAHA.117.008094. PMID 29754124
- See also: open access article from national library of medicine — https://pubmed.ncbi.nlm.nih.gov/29754124/